CLINICAL TRIAL: NCT06265571
Title: The Effect of Ultrasound-Guided Suprascapular Block Plus Low-dose Interscalen Brachial Plexus Block for Postoperative Pain in Shoulder Surgery
Brief Title: Postoperative Pain in Shoulder Surgery
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Ferda YAMAN, Principal Investigator, Eskisehir Osmangazi University
Other Study IDs: EskisehirUO
Record Dates: First submitted 2023-09-11; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GROUP I: Interscalene block (group I)15 ml of 0.5% bupivacaine was applied with a single injection to 12 of 18 patients,
  Interventions: Other: perineural injection
- GROUP II: 7.5 ml of interscalene and 7.5 ml of suprascapular block (GROUP II) were applied to 6 patients with posterior approach.
  Interventions: Other: perineural injection

INTERVENTIONS:
Other: perineural injection — perineural injection of local anesthestetic for postoperative pain management

SUMMARY:
After the approval of the ethics committee, the files of the patients who underwent arthroscopic shoulder surgery between 01.01.2019 and 01.03.2020 were evaluated retrospectively.

Data were recorded including age, gender, duration of anesthesia, duration of surgery, postoperative analgesia consumption, complications such as respiratory distress due to hemidiaphragmatic paralysis and complications such as hematoma and nerve damage due to block intervention.

DETAILED DESCRIPTION:
Patients who underwent arthroscopic shoulder surgery and underwent USG-guided interscalene block and concomitant suprascapular block were included in the study. We tried to determine whether there is a difference between different dose regimens in order to determine the effective analgesic dose and minimize the side effects of dose-dependent interscalene block applications.

ELIGIBILITY:
Inclusion Criteria:

arthroscopic shoulder surgery full data form

Exclusion Criteria:

chronic obstructive lung disease chronic opoid consumption missing data from the postoperative pain form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: >18 years old patients undergoing arthroscopic shoulder surgery by the same surgeon.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
rescue analgesia | between 01.01.2019 and 01.03.2020
  postoperative pain score (VAS) > 4 required to rescue analgesia
difference between the analgesic methods | between 01.01.2019 and 01.03.2020

CONTACTS AND LOCATIONS:
Overall Officials: Ferda YAMAN, Assoc prof, Study Director — University of Eskişehir Osmangazi
Locations (1):
- Ferda YAMAN, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
reterospectively completed